CLINICAL TRIAL: NCT05499195
Title: Selective Adjuvant Radiotherapy for pT1b Esophageal Cancer After Submucosal Endoscopic Resection- a Multicenter, Retrospective Study
Brief Title: Adjuvant Radiotherapy for pT1b Esophageal Cancer After Submucosal Endoscopic Resection
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhouguang Hui, M.D., Chief physician, Director of VIP Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC2690
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Cancer
Keywords: early-stage; submucosal endoscopic resection; adjuvant radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESD group: ESD was performed by a highly experienced endoscopist who underwent systemic training. First, the endoscopist carried out chromoendoscopy by spraying 1.25% Lugol's iodine solution to identify the lesion and made dots with a dual-knife outside the margin of the lesion. Next, a forward-viewing endoscope was introduced with a transparent cap attachment on its tip. A saline solution with methylene blue and epinephrine was injected into the submucosa with an injection needle to create a liquid cushion separating the lesion and the muscle layer. Then, a mucosal incision at the periphery of the marking dots was performed with a dual-knife. After that, the submucosal connective tissue beneath the lesion was dissected using the same dual-knife, and the lesion was totally removed through dissection.
- ESD+adjuvant radiotherapy group: The process of ESD was the same as that of ESD group. A total dose of 41.4-60.0 Gy in common fractionation based on three-dimensional conformal radiotherapy or intensity modulated radiotherapy technology was prescribed.

SUMMARY:
Endoscopic Resection (ER) is a crucial therapeutic and diagnostic method for superficial esophageal cancer. However, lymph node metastasis rate in pT1b patients is relatively high. Although, adjuavnt chemoradiotherapy is recommended, limied studies prove the superiority of additional adjuvant radiotherapy over ESD alone. This study aimed to further verify the efficacy of adjuvant radiotherapy in early-stage esophageal cancer after ESD.

DETAILED DESCRIPTION:
The incidence of early-stage esophageal cancer (EC) is increasing rapidly and even accounting for approximately 40% of esophageal squamous cell carcinoma. Endoscopic Resection (ER) is a crucial therapeutic and diagnostic method for superficial esophageal cancer. However, lymph node metastasis rate in pT1b patients is relatively high, and additional treatment is recommended after ER.

Adjuvant chemoradiotherapy is a treatment option and has already been proven to be equivalent to radical surgery. However, limited studies, with relatively small sample size and nature of low-level evidence, consistently showed that additional adjuvant radiotherapy failed to improve survival. Hence, adjuvant radiotherapy should not be applied without selection.

T1b EC patients are a heterogeneous population, with reported regional metastasis or recurrence rates varying considerably from 0-53% in SM1 disease, 19-31% in SM2, and 36-61% in SM3. The risk factors of regional metastasis or recurrence were also reported, generally including lymphovascular invasion (LVI) and pT1b disease.

In view of the aforementioned evidence, we hypothesized that selective adjuvant radiotherapy based on risk factors might significantly improve survival. The aim of this study was to evaluate the efficacy of adjuvant radiotherapy after ESD for pT1b EC and further explore the potential population who could benefit.

ELIGIBILITY:
Inclusion Criteria:

(1) ECOG score < 2; (2) Pathologically confirmed squamous or adenosquamous cell cancer; (3) Clinical stage cTis-1bN0M0; (4) Multiple primary T1 lesions were allowed; (5) No lymph nodes and distant metastases confirmed by chest CT, neck CT or neck ultrasound, and abdominal CT or abdominal ultrasound; (6) Underwent ESD between January 2010 and December 2019; (7) pT1b disease confirmed by endoscopically resected specimen; (8) Underwent adjuvant radiotherapy (with or without chemotherapy) or surveillance after ESD.

Exclusion Criteria:

(1) Diagnosed with other locally-advanced or advanced malignancies within 3 years before ESD; (2) Underwent radical surgery after ESD; (3) Upfront radiotherapy, chemotherapy or chemoradiotherapy before ESD; (4) Lost to follow-up or insufficient clinical information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who met the inclusion and exclusion Criteria treated in 11 hospitals in China were included.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3-year
  OS was defined as the duration between diagnosis and any cause of death.
Disease-free Survival (DFS) | 3-year
  DFS was defined as the duration between the diagnosis and any disease recurrence or any cause of death, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No